CLINICAL TRIAL: NCT03497481
Title: Appreciation of the Possibility of Dosing Neopterin in Eye Liquids. Pilot Study of Neopterin Dosage in Eye Liquids.
Brief Title: Neopterin Dosage in the Eye
Acronym: CHA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CHITS-02; 2017-A00183-47 (Other: Id-RCB)
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cataract
Keywords: eye's anterior chamber fluid; cerebrospinal fluid; inflammatory pathology
MeSH Terms: conditions — Cataract | interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — eye's anterior chamber fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neopterin Dosage: Eye's anterior chamber fluid and urines are sampled for posterior neopterin analysis
  Interventions: Biological: Samples

INTERVENTIONS:
Biological: Samples — Eye's anterior chamber fluid and urines are sampled for posterior neopterin analysis

SUMMARY:
The purpose of the study is to determine whether neopterin can be dosed in the fluid of the eye's anterior chamber for patient with non-inflammatory and non-infectious ophthalmic pathology.

DETAILED DESCRIPTION:
The study will be explained to subjects who are about to undergo ophthalmologic surgery. They will sign an informed consent and be included in the study. Urine sample will be collected specifically for the study. Eye's anterior chamber fluid will also be collected during the surgery as it is the usual practice (the sample is used for the neopterin dosage instead of being thrown away).

These samples will be centrifuged, frozen in a -80° C freezer. At the end of the study, all the samples will be sent to the central Lab for the neopterin dosage analysis. Results will be communicated to the principal investigator afterward.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old
* Non inflammatory or non infectious ophthalmic pathology requiring puncture of eye's anterior chamber fluid.
* Minimum of 200 microliter sample
* Immunocompetent subjects
* Signed and dated informed consent
* Samples management in accordance with the pre-analytical conditions specified in the protocol

Non-inclusion criteria:

* Age < 18 years-old
* Subjects treated with intraocular corticoids, antibiotics or anti-inflammatory, locally or in systemic injection, prior to inclusion.

Exclusion Criteria:

* Subjects who exercised his right of withdrawal
* Study suspended on principal investigator, sponsor or health authorities' demand.
* Deceased subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible for non infectious and non inflammatory eye surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Detection and dosage of neopterin in the eye | 3 month
  HCL will detect and dose the neopterin in the eye's anterior chamber fluid

SECONDARY OUTCOMES:
Neopterin concentration comparison between study values and reference value. | 3 month
  The reference values are standards established by the Neurobiology Lab from Lyon CHU which is the central lab that will performed the neopterin dosages.
False positives identification and elimination. | 3 month
  False positives will be determined by calibration of creatinine dosage in eye and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Chaker Nefzaoui, doctor, Principal Investigator — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer; Anélia Benarrosh, doctor, Study Chair — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Result] Kuvbachieva-Benarrosh A, Nefzaoui C, Quadrio I, Remignon CH, Jullian E, Perret-Liaudet A. Neopterin level can be measured by intraocular liquid biopsy. Clin Chem Lab Med. 2022 Oct 14;61(1):e20-e21. doi: 10.1515/cclm-2022-0691. Print 2023 Jan 27. No abstract available. PMID 36227583